CLINICAL TRIAL: NCT07124195
Title: A Randomized, Controlled, Multicenter Clinical Study on the Whole-Process Management of Nanocrystalline Megestrol in Preventing Chemotherapy-Induced Nausea and Vomiting
Brief Title: Nanocrystalline Megestrol for Managing Chemotherapy-Induced Nausea and Vomiting
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHASE012
Record Dates: First submitted 2025-08-02; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Malignant Solid Tumors; Moderate to High Emetogenic Chemotherapy (MEC/HEC) Drugs

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control-revention of CINV induced by HEC chemotherapy drugs (Other): Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily), Fosaprepitant (administered on Day 1, 150 mg, once daily)
  Interventions: Combination Product: high antiemetic regimen
- Control-Prevention of CINV induced by MEC chemotherapy drugs (Other): Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily)
  Interventions: Combination Product: moderate antiemetic regimen
- Prevention of CINV induced by HEC chemotherapy drugs (Experimental)
  Interventions: Drug: Medroxyprogesterone acetate oral suspension; Combination Product: high antiemetic regimen
- Prevention of CINV induced by MEC chemotherapy drugs (Experimental)
  Interventions: Drug: Medroxyprogesterone acetate oral suspension; Combination Product: moderate antiemetic regimen

INTERVENTIONS:
Drug: Medroxyprogesterone acetate oral suspension — Medroxyprogesterone acetate oral suspension (Meishiya®) (administered from Day 1 to 21, 5 ml, once daily)
  Arms: Prevention of CINV induced by HEC chemotherapy drugs; Prevention of CINV induced by MEC chemotherapy drugs
Combination Product: high antiemetic regimen — Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily), Fosaprepitant (administered on Day 1, 150 mg, once daily)
  Arms: Control-revention of CINV induced by HEC chemotherapy drugs; Prevention of CINV induced by HEC chemotherapy drugs
Combination Product: moderate antiemetic regimen — Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily)
  Arms: Control-Prevention of CINV induced by MEC chemotherapy drugs; Prevention of CINV induced by MEC chemotherapy drugs

SUMMARY:
The goal of this clinical trial is to learn if medroxyprogesterone acetate oral suspension (Meishiya®) works to prevent nausea and vomiting caused by single-day moderate to high emetogenic chemotherapy (MEC/HEC) in the whole-process management. It will also learn about the safety of medroxyprogesterone acetate oral suspension (Meishiya®). The main questions it aims to answer are:

Does medroxyprogesterone acetate oral suspension (Meishiya®) effectively prevent nausea and vomiting induced by single-day MEC/HEC in the whole-process management? What medical problems do participants have when taking medroxyprogesterone acetate oral suspension (Meishiya®)? Researchers will adopt a multicenter, randomized controlled, open-label trial design and compare the effects of medroxyprogesterone acetate oral suspension (Meishiya®) in preventing chemotherapy-induced nausea and vomiting.

Participants will be:

Stratified based on chemotherapy regimens (HEC vs MEC), gender (male vs female), and age (<55 years vs ≥55 years) Planned to be 126 subjects who are first-time recipients of single-day MEC/HEC for malignant solid tumors Take medroxyprogesterone acetate oral suspension (Meishiya®) as per the study protocol during the chemotherapy period Visit the research centers at specified intervals for checkups and assessments Record details of nausea, vomiting episodes, and any adverse reactions in a diary

DETAILED DESCRIPTION:
A Randomized, Controlled, Multicenter Clinical Study on the Whole-Process Management of Nanocrystalline Megestrol in Preventing Chemotherapy-Induced Nausea and Vomiting This study enrolls subjects with malignant solid tumors who are initially planned to receive moderate to high emetogenic chemotherapy (MEC/HEC) drugs. It aims to explore the efficacy and safety of medroxyprogesterone acetate oral suspension (Meishiya®) in the whole-process management of preventing nausea and vomiting caused by single-day moderate to high emetogenic chemotherapy (MEC/HEC) drugs. The study adopts a multicenter, randomized controlled, open-label trial design, with a planned enrollment of 126 subjects. Enrolled subjects will be stratified based on the following factors: chemotherapy regimens (HEC vs MEC), gender (male vs female), and age (<55 years vs ≥55 years).

The main interventions are as follows:

Prevention of CINV induced by HEC chemotherapy drugs (Cycles 1-2):

Experimental group: Medroxyprogesterone acetate oral suspension (Meishiya®) (administered from Day 1 to 21, 5 ml, once daily), Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily), Fosaprepitant (administered on Day 1, 150 mg, once daily) Control group: Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily), Fosaprepitant (administered on Day 1, 150 mg, once daily)

Prevention of CINV induced by MEC chemotherapy drugs (Cycles 1-2):

Experimental group: Medroxyprogesterone acetate oral suspension (Meishiya®) (administered from Day 1 to 21, 5 ml, once daily), Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily) Control group: Ondansetron Injection (administered on Day 1, 8 mg, once daily), Dexamethasone Tablets (administered on Day 1, 12 mg, once daily; administered from Day 2 to 4, 3.75 mg, twice daily) The trial consists of a screening period, a treatment period, and a safety follow-up period. Eligible subjects after screening will be randomly assigned to the experimental group or the control group in a 1:1 ratio, receive drug treatment according to the trial protocol, and then complete corresponding follow-ups and examinations in accordance with the trial flow chart. During the study, if the researcher assesses that the subject really needs to use rescue antiemetic drugs, rescue treatment can be carried out according to clinical practice. The specific type, usage, dosage, and frequency of the drugs will be determined by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years, regardless of gender;
* Histologically or cytologically confirmed malignant solid tumor;
* No prior exposure to any chemotherapy drugs (antitumor drugs not used for cancer treatment, or intravesical instillation therapy for bladder cancer is not considered as chemotherapy);
* Initially planned to receive single-day moderate to high emetogenic chemotherapy (MEC/HEC) drugs;
* Expected survival period ≥ 6 months;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Good organ function, meeting the following criteria:

  1. Neutrophil count ≥ 1.5×10⁹/L;
  2. Hemoglobin ≥ 90 g/L;
  3. Platelet count ≥ 100×10⁹/L;
  4. Total bilirubin ≤ 1.5×ULN;
  5. In patients without known liver metastasis, aspartate aminotransferase ≤ 2.5×ULN and/or alanine aminotransferase ≤ 2.5×ULN (for patients with liver metastasis, it can be relaxed to ≤ 5×ULN);
  6. Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 50 ml/min;
  7. Electrocardiogram: QTc ≤ 450 ms (male), QTc ≤ 470 ms (female);
  8. Echocardiogram: LVEF (left ventricular ejection fraction) ≥ 50%;
* Female subjects of childbearing potential and male subjects whose partners are female of childbearing potential need to use a highly effective contraceptive method from the time of signing the informed consent form until 6 months after the last dose (see Appendix VII); female subjects of childbearing potential must have a negative blood pregnancy test within 72 hours before randomization; and must be non-lactating;
* Clearly understand and voluntarily participate in the study, and sign the informed consent form in person.

Exclusion Criteria:

* Having received abdominal (including the diaphragmatic plane and below) or pelvic radiotherapy within 7 days before enrollment, or planning to receive such radiotherapy within days 1 to 8 of treatment;
* Planning to receive other moderate to high emetogenic chemotherapy drugs within days 2 to 8 after the first day of chemotherapy;
* Planning to receive chemotherapy regimens including conventional paclitaxel (using castor oil as solvent);
* Having taken drugs with potential antiemetic effects within 2 days before enrollment: 5-HT3 receptor antagonists (e.g., ondansetron, etc.), phenothiazines (e.g., prochlorperazine), butyrophenones (e.g., haloperidol), benzamides (e.g., metoclopramide), domperidone, cannabinoids, traditional Chinese medicines with potential antiemetic effects, scopolamine, cyclizine, etc.;
* Having started treatment with benzodiazepines or opioids within 2 days before enrollment (except for triazolam, temazepam or midazolam taken alone daily);
* Subjects who started using morphine within 7 days before enrollment (except those taking a stable dose);
* Having received systemic corticosteroid therapy (including but not limited to dexamethasone, hydrocortisone, methylprednisolone or prednisolone) or sedative antihistamines (such as diphenhydramine) within 7 days before enrollment (Note: single use of steroids to prevent contrast agent allergy and local or inhaled administration are allowed);
* Having used palonosetron within 14 days before enrollment;
* Having used NK-1 receptor antagonists within 28 days before enrollment;
* Having used specific CYP3A4 substrates (terfenadine, cisapride, astemizole) or CYP3A4 inhibitors (such as ritonavir, clarithromycin, ketoconazole or itraconazole, diltiazem, etc.) within 7 days before enrollment, and having used strong CYP3A4 inducers (such as phenobarbital, rifampicin, phenytoin and carbamazepine, etc.) or specific CYP2D6 substrates (thioridazine, pimozide) within 28 days before enrollment;
* Having vomiting and/or retching, nausea within 24 hours before enrollment;
* Subjects with symptomatic brain metastasis or any symptoms suggesting brain metastasis or intracranial hypertension;
* Accompanied by poorly controlled serous cavity effusions, including pleural effusion, ascites, pericardial effusion (those controlled after treatment and stable for ≥ 2 weeks can be included);
* Having severe cardiovascular diseases within 3 months before enrollment, including but not limited to acute myocardial infarction, unstable angina pectoris, significant valvular or pericardial diseases, history of ventricular tachycardia, symptomatic chronic heart failure (New York Heart Association [NYHA] class II to IV), history of severe cardiac conduction abnormalities (such as torsades de pointes);
* Having poorly controlled hypertension before enrollment (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at two consecutive resting measurements);
* Complicated with active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10⁴ copies/mL), active hepatitis C (HCV-Ab positive, and HCV-RNA ≥ upper limit of normal), acquired immunodeficiency syndrome (AIDS) or positive HIV test, positive syphilis test;
* Complicated with concomitant diseases that cannot take dexamethasone, such as active infection (e.g., pneumonia) or any uncontrolled diseases (e.g., diabetic ketoacidosis, gastrointestinal obstruction, etc.);
* Known contraindications to NK-1 receptor antagonists, 5-HT3 receptor antagonists or dexamethasone; history of thromboembolic diseases within the past 6 months;
* Having participated in other clinical trials within 30 days before enrollment (based on the use of study drugs);
* Subjects considered by the researcher to be unsuitable for participating in this study due to other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the efficacy of medroxyprogesterone acetate oral suspension (Meishiya®) in the whole-process management of preventing nausea and vomiting induced by single-day moderate to high emetogenic chemotherapy (MEC/HEC) drugs. | 42 days
  The proportion of patients with no nausea during the entire period (Day 1 to Day 21) after the start of chemotherapy administration in the first chemotherapy cycle.

SECONDARY OUTCOMES:
the safety of medroxyprogesterone acetate oral suspension (Meishiya®) in the whole-process management of preventing nausea and vomiting induced by single-day moderate to high emetogenic chemotherapy (MEC/HEC) drugs. | 42 days
  The proportion of patients with any kind of adverse effects.
Quality of life score assessed by FLIE scale | 42 days
  Quality of life assessed by Functional Living Index-Emesis (FLIE). The FLIE scale ranges from 0 to 108, with higher scores indicating better quality of life (less impact of emesis on daily functioning)
Quality of life score assessed by EORTC QLQ-C30 | 42 days
  Quality of life assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). This questionnaire includes functional scales (range: 0-100; higher scores indicate better physical/role/emotional functioning) and symptom scales (range: 0-100; higher scores indicate more severe symptoms such as fatigue or pain).
Quality of life score assessed by EQ-5D scale | 42 days
  Quality of life assessed by EuroQol 5-Dimension Questionnaire (EQ-5D). The EQ-5D index score ranges from -0.594 to 1 (in general population norms), with higher scores indicating better health-related quality of life.

OTHER OUTCOMES:
Cytokine levels in blood | 42 days
  Levels of cytokines in blood samples, measured by detecting differences in proteomic expression from blood samples collected before medication.
Occurrence of nausea and vomiting after treatment | 42 days
  Incidence and severity of nausea and vomiting in patients after treatment, analyzed in association with proteomic factors (from pre-medication blood samples).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China